CLINICAL TRIAL: NCT00690001
Title: The Detection of Drug-Resistant HIV-1 in Taiwan
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Szu-Min Hsieh, National Taiwan University Hospital
Other Study IDs: 200803084R
Record Dates: First submitted 2008-06-01; First posted 2008-06-04 (Estimated); Last update posted 2008-07-08 (Estimated); Status verified 2008-04

CONDITIONS: HIV Infections
Keywords: HIV-1 infection; Treatment Experienced
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: HIV-1 infected patients in Taiwan

SUMMARY:
To assess the HIV resistance rate to variable antiretroviral agents in Taiwan, especially in patients with treatment failure, and to know the correlation between the drug resistance pattern and the HIV subtype, we will enroll a total of 150~200 HIV-1-infected subjects to perform genotypic resistance testing and try to establish facility of phenotypic resistance testing.

DETAILED DESCRIPTION:
Drug-resistant HIV strains may develop during antiretroviral therapy, and transmission of drug-resistant virus has been documented to be possible. The emergence of drug resistance in HIV has been associated with suboptimal virologic response to antiretroviral therapy [1]. The likelihood that a patient will acquire drug-resistant virus is related to the prevalence of drug resistance in the population with specific high-risk behaviors. In the western countries, studies suggest that the prevalence of viral resistance to at least one antiretroviral drug ranges from 6% to 16% in treatment-naïve patients, and among them, about 3% to 5% with reduced susceptibility to more than one class [2-4]. However, there is no data addressing the prevalence of drug resistance in various populations in Taiwan currently.

Drug resistance can be measured using either genotypic or phenotypic resistance assays. Genotypic assays detect mutations that cause dug resistance; phenotypic assays are drug susceptibility assays that measuring the in vitro ability of the virus to grow in the presence of serial dilutions of the inhibitors (that is, antiretroviral drugs). Because of its more rapid turnaround time and less expensiveness, a genotypic assay is generally preferred to phenotypic assay [5]. Genotypic resistance assay has been available in three AIDS centers in Taiwan. However, the methods used for genotypic assay are different in the three centers, and these data have not been gathered and analyzed to know the epidemiology of HIV resistance in Taiwan, thus the interpretation and application of the results from genotypic resistance assay for selection of antiretrovirals are quite questionable in Taiwan.

Furthermore, though the genotypic assay is less straightforward, several conditions exist to cause the discordance between genotype and phenotype, and the discordance may result in the difficulty in phenotype prediction from genotype [6]. Thus, phenotypic assay may help interpretation of resistance testing results and provide a guide to decide the optimal regimen. With the availability of newer classes of antiretrovirals in the near future, currently commercially available phenotypic testing using the recombinant viruses with insertion of reverse transcriptase and protease gene sequences may not be enough. A new phenotypic assay that can measure the virus ability to grow in the different concentrations of NRTIs, NNRTIs, PIs, entry inhibitors, CCR5 inhibitors and integrase inhibitors will be needed.

It has been known that HIV-1 load in plasma is strongly correlated with disease progression, response to antiviral treatment, and transmission from mother to child. The plasma viral RNA is more representative of the replicating virus pool at any time point than the cell-associated proviral DNA. In order to study the relationship of the complete HIV-1 genome to phenotypic resistance, we choose to focus on plasma virions. However, for those patients whose plasma viral load is not high enough to conduct this analysis, we will instead of using patients' proviral DNA from infected PBMC for phenotypic resistance analysis. Two strategies will be used to amplify viral genome. The first one will be amplification of a nearly full-length viral genome. If this strategy does not work, the second strategy will be to amplify two fragments of viral genome and to assemble these two fragments by unique restriction enzymes.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1-infected subjects under antiretroviral therapy if they are 20 ~ 60 years old and have a plasma HIV RNA > 1000 copies/mL and give inform consents will be enrolled.

Exclusion Criteria:

* with antiretroviral therapy within 4 weeks

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: HIV-1-infected patients under antiretroviral therapy with clinical suspicion of emergence of virus resistance
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2008-04

PRIMARY OUTCOMES:
genotypic resistance testing | May 2009

CONTACTS AND LOCATIONS:
Overall Officials: Szu-Min Hsieh, M.D., Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan